CLINICAL TRIAL: NCT05825534
Title: Pressure Opening With Electrical Impedance Tomography
Acronym: POET
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Collaborators: Unity Health Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: PI2022_843_0159
Record Dates: First submitted 2023-04-11; First posted 2023-04-24 (Actual); Last update posted 2023-09-13 (Actual); Status verified 2023-09

CONDITIONS: Acute Respiratory Distress Syndrome; Acute Lung Injury
Keywords: airway closure; airway opening pressure; Acute Respiratory Distress Syndrome; Acute Lung Injury
MeSH Terms: conditions — Respiratory Distress Syndrome; Acute Lung Injury

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- EIT monitoring (Experimental)
  Interventions: Other: EIT monitoring

INTERVENTIONS:
Other: EIT monitoring — EIT monitoring (PulmoVista 500, Dräger, Lübeck, Germany) will be applied using a dedicated silicon belt with 16 electrodes placed at the level of the fifth intercostal space. The EIT system will be connected to the ventilator and data of gas flow, volume, airway pressure, and impedance will be synchronously collected at 40 Hz. The investigators will perform one simple pressure-volume (PV) curve with a low-flow insufflation of 5 L/min starting from 0 cmH2O. During the low-flow insufflation, both ventilator and EIT-derived PV curves will be recorded. All PV curves will be analysed offline to detect complete and regional airway closures, and measure AOPs.

SUMMARY:
Acute lung injury and ARDS (acute respiratory distress syndrome) are characterized by lung inhomogeneity, leading to a different distribution of the tidal volume (and pressure) within the lung. The quasi-static PV curve is a useful bedside tool to set mechanical ventilation, but it reflects a global behaviour of the lung. The electrical impedance tomography (EIT) is a non-invasive and radiation-free tool, monitoring dynamic changes in gas distribution. Images from EIT can be divided in several regions of interest, allowing to measure regional changes in compliance. The regional derived-EIT PV curve could provide valuable information on airway closure and AOP (airway opening pressure). Recent studies suggest that AOP measured by the ventilator seems to correspond to the AOP of the lowest injured lung. The investigators will perform one pressure-volume (PV) curve with a low-flow insufflation of 5 L/min starting from 0 cmH2O to a maximal airway pressure corresponding to the plateau pressure. During the low-flow insufflation, both ventilator and EIT-derived PV curves will be recorded. All PV curves will be analysed offline by the investigator to detect complete and regional airway closures, and measure AOPs.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (≥18 years old).
* Patients with PaO2/FiO2 ratio <300 mmHg.
* Volume- or pressure-controlled ventilation.
* Sedated, with or without infusion of neuromuscular blockage.
* Patients in supine position

Exclusion Criteria:

* Pneumothorax and bronchopleural fistula.
* Severe hemodynamic instability (>30 % increase in vasopressors in the last 6 hours or norepinephrine > 0.5 µg/kg/min).
* PaO2/FiO2 ratio < 80 mmHg.
* Severe or very severe chronic obstructive pulmonary disease (COPD) according to the GOLD criteria (stage III: FEV1 30-50% predicted; stage IV: FEV1 < 30 % predicted).
* Known or highly suspected elevated intracranial pressure (>18 mmHg).
* Impossibility to correctly position the EIT belt (e.g., burns chest drainage, etc.).
* Contraindications to EIT (e.g., implantable cardiac defibrillator, pacemaker, instable spinal lesions, etc.).
* Clinical judgement of the attending physician.
* Pregnant or breastfeeding woman
* Patient under guardianship, curators or safeguard of justice

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-06-23 (Actual); Primary Completion 2024-05 (Estimated); Study Completion 2024-05 (Estimated)

PRIMARY OUTCOMES:
prevalence of regional airway closure | 1 year
prevalence of complete airway closure | 1 year
Difference of global AOP values between EIT-derived method and the highest regional AOP | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHU Amiens, Amiens, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sun N, Brault C, Rodrigues A, Ko M, Vieira F, Phoophiboon V, Slama M, Chen L, Brochard L. Distribution of airway pressure opening in the lungs measured with electrical impedance tomography (POET): a prospective physiological study. Crit Care. 2025 Jan 16;29(1):28. doi: 10.1186/s13054-025-05264-3. PMID 39819779